CLINICAL TRIAL: NCT03184779
Title: Ski and Snowboard School Programs: Assessing the Effect of a Safety Video Intervention on Knowledge, Behaviour and Injury Risk in Youth Skiing and Snowboarding
Brief Title: The Effect of a Safety Video on Ski and Snowboard School Program Participants in Calgary, Alberta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sport Injury Prevention Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB15-0749
Record Dates: First submitted 2017-05-02; First posted 2017-06-14 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-04

CONDITIONS: Knowledge, Attitudes, Practice; Risk Behavior; Injuries
Keywords: Ski; Snowboard; Snow Sport; Injury; Injury Prevention; Safety; Safety Video; Video Intervention; Youth; Children; Adolescent; Education; Knowledge
MeSH Terms: conditions — Behavior; Risk-Taking; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Schools will be stratified by grade and half of the schools in each stratum will be randomly assigned to the intervention and the other half will be assigned to the control group. Stratification by grade is necessary to ensure that groups are similar enough to ensure less biased comparisons. The research team will also ensure that schools going on their outing to COP on the same day are assigned to the same group. This is to ensure that research assistants can assume that all students observed on the hill for that particular day have the same intervention or control status since it may be challenging to distinguish which school group each student belongs to strictly through observation. That way the research team can accurately ascertain the intervention and control status of each student for the behavior observation component of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants (including the teachers and students) will not be told by the research team if the video assigned to their class is the control or intervention. During the consent process though, they will be made aware that they are going to be randomly assigned to either the control or intervention video.
  Furthermore, when the two observers go to the ski hill to collect data on observed unsafe behaviours, they will be blinded to the intervention/control status of the school at the ski area that day to prevent observer bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive an educational video containing safety messages and an injury prevention component with the intent of reducing behaviours and actions on the hill than can potentially lead to injury.
  Interventions: Other: Ski and Snowboard Safety Video
- Control (No Intervention): The control group will receive the usual procedures associated with school outings where students have the opportunity to watch the standard welcome video (~8 minutes) with information on how their day will go and how to use and put on safety equipment. The information given in the control procedure emphasizes preparation and how to use and put on equipment rather than safety messages oriented towards preventing injury and collisions. Students in the control group will watch the video prior to participating in the ski area school program.

INTERVENTIONS:
Other: Ski and Snowboard Safety Video — The ski and snowboard safety video (~10 minutes) includes information on preparation, correct protective equipment use (e.g. helmets), and strategies for speed control and collision avoidance. Focus groups were conducted among parents, students, ski patrol, and ski instructors to inform the content and format of the video. Feedback and suggestions from focus groups were utilized to ensure that the video optimized information uptake from children and adolescents who watch the video. The Health Action Process Approach (HAPA) model was embedded throughout the video to ensure evidence-informed pathways towards positive behaviour change.
  Arms: Intervention

SUMMARY:
The main objective of the study is to investigate if a video intervention can help increase knowledge, decrease risky behaviours on the hill, and reduce injury risk in students who participate in ski and snowboard school programs. The study design is a cluster randomized controlled trial where participating schools will be randomized into either an intervention or control group. The intervention video will contain an injury prevention and safety promotion component for skiing or snowboarding. The control group will receive the standard orientation video that many schools typically provide for students prior to their ski/snowboard outings in previous years.

DETAILED DESCRIPTION:
Skiing and snowboarding are two popular winter activities, and school sanctioned ski and snowboard programs hosted at local ski areas provide students the opportunity to discover and engage in new activities that can benefit their physical and mental well-being. However, these winter sports can be associated with a high risk of injury. Previous studies have found that the majority of injuries in snow sports are preventable and tend to be caused by poor decisions, actions and human error. As part of ski and snowboard school programs at WinSport's Canada Olympic Park (COP) in Calgary, Alberta, children receive an introduction to the sport including basic safety information. However, there is no consistent and comprehensive injury prevention component built into ski and snowboard school outing programs. For this research, the investigative team will implement and evaluate a video intervention with built-in injury prevention and safety promotion messages.

The study design is a cluster randomized controlled trial where participating schools will be randomized into either an intervention or control group. The intervention video is approximately 10 minutes in length and will include information on proper preparation, correct protective equipment use, and strategies for speed control and collision avoidance while skiing or snowboarding. The content and format of the intervention video was developed and informed by focus groups with parents, students, ski patrollers, and ski instructors to ensure optimal information uptake for viewers.The control group will receive the standard orientation video that many schools usually provide for students prior to their ski/snowboard outings.

The participants will be children between the ages of 6 to 15 years (grades 1 to 9) who participate in the ski and snowboard school programs at COP in Calgary, Alberta. The outcomes of interest that will be measured include knowledge uptake (through the use of pre- and post-test questionnaires delivered before and after watching the assigned video, and measuring differences in test scores before and after watching the video), behavioural changes (through the use of multiple observers who will collect data on unsafe behaviours and actions observed on the ski hill during two hour time intervals) and injury risk (through the use of nationally standardized ski patrol accident report forms that will be provided by the ski area and school program enrollment data to calculate injury rates).

ELIGIBILITY:
Inclusion Criteria:

* Elementary and junior high school students (grades 1 to 9)
* Attends a school participating in a ski and snowboard school program hosted by a local ski area

Exclusion Criteria:

* High school students (grade 10 or above)

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2348 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge Uptake | Throughout the ski/snowboard season (up to 5 months)
  Students will take a baseline safety knowledge assessment before watching the assigned video (pre-test) and take the same test immediately after watching the assigned video (post-test). The video viewing and the pre- and post-test completion will be moderated in a classroom by the teacher and a member of the research team. Questions about preparations, equipment and proper hill etiquette will be included in the knowledge assessment questionnaire.
  At the start of the data collection session at the school, demographic information will be collected followed by the pre-test knowledge assessment for students to complete independently. After the pre-test knowledge assessment is completed and submitted, the students will then watch their assigned video. Immediately following the video, the students will independently complete the post-test knowledge assessment. A follow-up assessment test will be given to the participants approximately 1 month after watching the video.

SECONDARY OUTCOMES:
Risky Behaviours | Throughout the ski/snowboard season (up to 5 months)
  Two research assistants (RAs) will observe the behaviour and characteristics of school participants during 2-hour intervals. Data will be collected on multiple unsafe behaviours, including: obstructing the run, stopping in an area where they are not visible, not yielding or giving right of way to skiers/snowboarders below, skiing/snowboarding too close to others, excessive speed, and jumping unsafely. RAs will select and agree on the next student who comes off the magic carpet to observe. When both observers are ready, they will give each other a cue and start observing the same student as they go down the hill. The RAs will stop observing and recording data on that student when the student reaches the bottom of the run. Once both RAs have recorded their data and confirm they are ready for the next student, they will choose the next student for observation. The number of students in the ski area during the time periods will also be recorded for denominator data as students per hour.
Injury | Throughout the ski/snowboard season (up to 5 months)
  Injury data will be obtained from the ski patrol Accident Report Forms (ARF). ARFs are completed by ski patrollers and contain information on the circumstances surrounding the injury, as well as the demographic characteristics of the injured skier or snowboarder. The forms also include information on whether those who were injured were participating in a school program at the time of injury. All personal identifying information will be removed from ARFs by ski patrol before being given to the research team for analysis. The name of the school and the date and time of the injury will be used to link ski patrol ARF injury data to the intervention or control schools. Denominator data will be the school program data; these data contain information on which schools were at the ski area for each day and the number of participants. This information is entered by school teachers and compiled by WinSport.

CONTACTS AND LOCATIONS:
Overall Officials: Brent E Hagel, PhD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: Undecided